CLINICAL TRIAL: NCT02651831
Title: Development and Validation of a Health-related Quality of Life Instrument: Functional Assessment of Cancer Therapy - Immune Checkpoint Modulators, an Investigator Initiated Study (FACT-ICM).
Brief Title: Development and Validation of a Health-related Quality of Life Instrument
Acronym: FACT-ICM
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: FACT-ICM
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: ICMs; Immune checkpoint modulators
MeSH Terms: conditions — Neoplasms | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1A: Content Validation: Up to 4 focus groups of 6-10 cancer patients each will be conducted each lasting approximately 90 mins. An additional 10 to 15 patients will undergo individual semi-structured interviews each lasting around 60 minutes.
  10-12 expert clinicians experienced in treating patients with ICMs or managing ICM toxicities will participate in a survey, and group or individual interviews.
  Interventions: Other: Focus groups and individual interviews
- 1B: Face Validity: Patients who have been and are being treated with ICMs to complete draft questionnaire (FACT-ICM). Some patients who were involved in the first round of interviews will be re-interviewed, and interview naïve patients will also be included.
  Interventions: Other: Questionnaire
- 2A: To measure test-retest reliability: Patients to complete FACT-ICM at at two time points separated by 5 to 14 days.
  Interventions: Other: Questionnaire
- 2B: To confirm construct validity: To evaluate discriminative properties of FACT-ICM, scores will be compared between pre-defined groups of patients where differences are expected.
  Interventions: Other: Questionnaire
- 2C: To determine responsiveness and MCID: Responsiveness testing: Patients will complete FACT-ICM within a week of starting treatment, then while on treatment and within 30 days after end of treatment (EOT) with ICMs.
  MCID testing: In addition to the FACT-ICM score, patients undergoing serial assessment for responsiveness will also indicate how much better or worse they are using a 5-point rating scale.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Focus groups and individual interviews — Focus groups conducted to explore general experiences, insights and concerns of those receiving ICM therapies. Individual semi-structured interviews to provide in-depth data on the themes identified in the focus groups.
  Groups: 1A: Content Validation
Other: Questionnaire — Health related quality of life questionnaire (FACT-ICM) to be completed by patients
  Groups: 1B: Face Validity; 2A: To measure test-retest reliability; 2B: To confirm construct validity; 2C: To determine responsiveness and MCID

SUMMARY:
This study aims to develop a health related quality of life (HRQOL) patient reported outcome (PRO) for patients receiving immune checkpoint modulator (ICM) therapy. This instrument could be used to in clinical trials to evaluate HRQOL for patients treated with novel ICMs and ICM combinations that might ultimately influence decisions about regulatory approval, as well as improved understanding of chronic treatment effects on patient well-being, understanding reasons for treatment non-adherence, and developing strategies to improve adherence and evaluating clinical outcomes.

DETAILED DESCRIPTION:
Immune Checkpoint Modulators (ICMs) are associated with significant adverse events. Currently there are no validated patient reported outcome (PRO) tools to assess health related quality of life (HRQOL) specifically in patients receiving ICMs. HRQOL is a multidimensional concept of a patient's perceived well-being that can be affected by disease and treatment. There is an urgent need to assess the impact of ICMs on HRQOL, to better understand the balance between efficacy and toxicity with these agents.

This study aims to develop a health related quality of life (HRQOL) patient reported outcome (PRO) for patients receiving immune checkpoint inhibitor (ICM) therapy (FACT-ICM). The core domains of the FACT-ICM will include physical, emotional, family and social, and functional well being. In addition, the proposed study will develop a toxicity sub-scale related to resultant toxicities from ICM therapy.

The HRQOL will be developed through focus groups and interviews with patients treated with ICMs, and clinicians treating patients with ICMs, to understand how treatment with ICMs impacts HRQOL, as well as explore general experiences, insights and concerns of those receiving ICM therapies.

ELIGIBILITY:
Inclusion Criteria:

Patient Criteria

* Cancer diagnosis (any type, advanced or metastatic stage);
* Treatment with an agent or agents that modulate an immune checkpoint (any line of therapy);
* Age ≥ 18;
* English-speaking;
* ECOG PS 0-3
* Able to complete questionnaires independently
* Able to provide informed consent.
* Completed treatment within a year of enrolment

Clinician Criteria

* Must either treat patients with ICMs or manage side effects of patients treated with ICMs
* Be able to attend interviews and participate in discussions as part of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be patients who are receiving treatment that modulates immune checkpoints and clinicians with expertise in this area.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2015-07; Primary Completion 2024-01 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
Confirmatory factor analysis of FACT-ICM PRO tool variables compared to content analysis and qualitative descriptives of patient focus groups and interviews in target group | 6 months

SECONDARY OUTCOMES:
Change of score for each domain and also the total FACT-ICM score at baseline to 5-14 days for patients with minimal change in status | 5-14 days
Comparison of FACT-ICM scores between pre-defined groups of patients where differences are expected | 6 months
FACT-ICM change scores from baseline to within 30 days after end of treatment | Baseline, an average of 3 months, and within 30 days after end of treatment
Change in MCID values from baseline to within 30 days after end of treatment | Baseline, an average of 3 months, and within 30 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada